CLINICAL TRIAL: NCT01588912
Title: A Randomized, Prospective, Multicenter, Open-label Study to Evaluate the Efficacy of Telbivudine With or Without add-on Tenofovir According to Roadmap Strategy Compare With Entecavir in HBeAg-positive Chronic Hepatitis B Patients
Brief Title: Efficacy of Telbivudine With or Without add-on Tenofovir According to Roadmap Strategy Compare With Entecavir
Acronym: TETRA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Ki Tae Yoon, Assistant Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600AKR07T
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B; HBeAg positive; telbivudine; tenofovir; entecavir; roadmap
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine; Tenofovir; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telbivudine-Tenofovir roadmap (Experimental)
  Interventions: Drug: Telbivudine; Drug: Tenofovir
- Entecavir (Active Comparator)
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Telbivudine — If virologic response, which means HBV DNA < 50 IU/mL, is shown at 24 weeks, telbivudine monotherapy is maintained and in the event that virologic response is not shown, tenofovir add-on therapy is done
  Other Names: Sebivo
  Arms: Telbivudine-Tenofovir roadmap
Drug: Tenofovir — If virologic response, which means HBV DNA < 50 IU/mL, is shown at 24 weeks, telbivudine monotherapy is maintained and in the event that virologic response is not shown, tenofovir add-on therapy is done
  Other Names: Viread
  Arms: Telbivudine-Tenofovir roadmap
Drug: Entecavir — Maintain the entecavir through the study period
  Other Names: Baraclude
  Arms: Entecavir

SUMMARY:
Oral antiviral drugs which can be given to patients with HBeAg-positive chronic hepatitis B include Lamivudine, Clevudine, Adefovir, Telbivudine, Entecavir and Tenofovir. 2009 American Association for the Study of Liver Disease (AASLD) Treatment Guidelines and 2009 European association for the Study of the Liver (EASL) Treatment Guidelines recommend the administration of Entecavir or Tenofovir with high potency and low resistance. Lamivudine has low antiviral potency and high incidence of mutation in long-term administration compared to Entecavir or Tenofovir. Clevudine causes the elevated creatinine kinase (CK), side effects including myositis/myopathy and much mutation in the long-term administration. Globe study demonstrated Telbivudine had more excellent antiviral potency than Lamivudine, which was also comparable to or higher than Entecavir or Tenofovir. Nevertheless, the choice of treatment drugs can be limited due to the mutation rate of 25% for 2 years. However, the analysis of Globe study results showed that 2-year treatment progress was very good in patient who showed virologic response at 24 weeks after the initiation of treatment and that high antiviral potency and low mutation rate were observed when the Telbivudine roadmap strategy (in the event that virologic response is shown at 24 weeks, telbivudine monotherapy is maintained and in the event that virologic response is not shown, tenofovir add-on therapy is done) recently implemented and announced in 2011 Asian Pacific Association for the Study of the Liver (APASL) was applied. However, the study was single arm study, which restricted the comparison between Entecavir and Tenofovir monotherapy groups. Therefore, this study intends to compare the anti-viral effect and mutation rate between Entecavir 0.5mg monotherapy group and Telbivudine roadmap strategy group in patients with HBeAg-positive chronic hepatitis B through a randomized study.

DETAILED DESCRIPTION:
104 treatment-naïve patients with HBeAg-positive chronic hepatitis B who fulfill the inclusion criteria will be randomized in a 1:1 ratio to receive either Telbivudine 600mg monotherapy or Entecavir monotherapy with stratification before randomization according to presence of cirrhosis. For Telbivudine group, Telbivudine monotherapy or Tenofovir combined therapy will be done according to virologic response at 24 weeks and the primary study will be completed at Week 48 and treatment response will be analyzed. The treatment will be extended to Week 96 and the secondary analysis will be performed then.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age
* Documented CHB defined by HBsAg or HBeAg positive at least 6 month prior
* HBsAg positive at screening visit
* HBeAg positive and Anti-HBe negative at screening visit
* Serum HBV DNA 20,000~200,000,000 IU/mL as determined by Realtime PCR at screening visit
* Serum ALT 80~400 IU/mL at screening visit
* Patient is willing and able to comply with the study drug regimen and all other study requirements
* Patient is willing and able to provide written informed consent to participate in the study

Exclusion Criteria:

* Patient has received interferon, pegylated interferon, nucleoside or nucleotide drugs at any time
* Patient is co-infected with HCV, HDV, or HIV
* Patient with Child Pugh B or C (Child Pugh score ≥ 7)
* Patient has a history of or clinical signs/symptoms of hepatic decompensation such as ascites, esophageal variceal bleeding, hepatic encephalopathy
* Patient has any of the following laboratory values at screening visit:
* Hemoglobin <10 g/dL
* Absolute neutrophil count (ANC) <1,500/mm3
* Platelet count <70,000/mm3
* Patient has a history of clinical and laboratory evidence of chronic renal insufficiency defined as an estimated serum creatinine clearance < 50 mL/min using the MDRD formula at screening visit
* Patient is pregnant or breastfeeding
* Patient with currently abusing illegal drugs or alcohol sufficient
* Patient has organ transplantation
* History of any other acute or chronic medical condition that in the opinion of the investigator would make the patient unsuitable for inclusion into the study
* Patient has one or more additional known primary or secondary causes of liver disease, other than CHB, including steatohepatitis and autoimmune hepatitis
* Patient, if AFP is >50ng/mL at screening visit, has image findings suggestive of HCC at Liver CT or Liver MRI
* Patient with hypersensitivity for study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
HBV DNA non-detectability | Week 48
  Low detection limit of HBV DNA is 50 IU/mL

SECONDARY OUTCOMES:
HBV DNA non-detectability | Week 96
  Low detection limit of HBV DNA is 50 IU/mL
Reduction of HBV DNA from baseline | Week 12, 24, 36, 48, 60, 72, 84 & 96
HBeAg loss or HBeAg seroconversion | Week 48 & 96
HBsAg loss or HBsAg seroconversion | Week 48 & 96
ALT normalization | Week 48 & 96
Accumulate rate of Viral breakthrough | Week 48 & 96
Accumulate rate of Biochemical Breakthrough | Week 48 & 96
Accumulate rate of genotypic mutation in HBV | Week 48 & 96
Change of eGFR from baseline | Week 12, 24, 36, 48, 60, 72, 84 & 96
Accumulate rate of CK abnormal elevation | Week 48 & 96
Accumulate rate of symptom related muscular disease | Week 48 & 96
Accumulate rate of Adverse event or serious adverse event | Week 48 & 96

CONTACTS AND LOCATIONS:
Overall Officials: Ki Tae Yoon, M.D., Principal Investigator — Pusan National University Yangsan Hospital
Locations (10):
- South Korea (10):
  - Byung Chul Yoon, Busan
  - Eun Uk Jung, Busan
  - Hyun Young Woo, Busan
  - Nae-Yun Heo, Busan
  - Yang Hyun Baek, Busan
  - Hyun Jin Jo, Changwon
  - Byung Seok Kim, Daegu
  - Soo Young Park, Daegu
  - Hyun Ju Min, Jinju
  - Ki Tae Yoon, Yangsan